CLINICAL TRIAL: NCT00002234
Title: A Phase II, 48 Week, Open-Label Study Designed to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of a Simplified Dosing Regimen of Preveon (Adefovir Dipivoxil; bis-POM PMEA), Videx (Didanosine; ddI), Sustiva (Efavirenz; DMP-266), and Epivir (Lamivudine; 3TC) Administered Once Daily for the Treatment of HIV-1 Infection
Brief Title: Safety and Effectiveness of Giving an Anti-HIV Drug Combination of Adefovir Dipivoxil Plus Didanosine Plus Efavirenz Plus Lamivudine Once Daily to HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry); Dupont Applied Biosciences (Industry)
Organization: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: 232J; ICC 604
Record Dates: First submitted 2001-08-30; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; adefovir dipivoxil; Lamivudine; Didanosine

INTERVENTIONS:
Drug: Efavirenz
Drug: Adefovir dipivoxil
Drug: Lamivudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give HIV-infected patients a new combination of anti-HIV drugs taken once daily.

DETAILED DESCRIPTION:
Patients receive a treatment regimen of adefovir dipivoxil, didanosine, efavirenz, and lamivudine for 48 weeks. During the study, patients are evaluated for changes from baseline in plasma HIV-1 RNA and lymphocyte subsets and for the development of adverse experiences and laboratory toxicities. At Weeks 8, 12, 24, and 48, patients are assessed for adherence to study treatment with a questionnaire. Patients who experience virologic failure are discontinued from the study. Patients who experience treatment intolerance may have their antiretroviral treatment regimens changed. After Week 48, patients with documented virologic response are eligible to continue receiving study treatment.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are at least 13 years old (need consent of parent or guardian if under 18).
* Have an HIV count of 5,000 copies/ml or more within 30 days prior to study entry.
* Have a CD4+ count of 50 cells/mm3 or more.

Exclusion Criteria

You will not be eligible for this study if you:

* Are diagnosed with hepatitis within 30 days prior to study entry.
* Have certain serious medical conditions, including an AIDS-defining clinical condition.
* Received chemotherapy or radiation therapy within 30 days of study entry.
* Have taken any nucleoside reverse transcriptase inhibitors (NRTIs) for more than 2 weeks.
* Have ever taken 3TC.
* Have ever taken any non-nucleoside reverse transcriptase inhibitors (NNRTIs).
* Have taken medications that affect your immune system within 30 days prior to study entry.
* Have received a vaccine within 30 days prior to study entry.
* Are enrolled in another anti-HIV drug study while participating in this study.
* Abuse alcohol or drugs.
* Are pregnant or breast-feeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pacific Oaks Med Group, Beverly Hills, California
  - Univ of Colorado / Health Science Ctr, Denver, Colorado
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Brown Univ School of Medicine, Providence, Rhode Island
  - Hampton Roads Med Specialists, Hampton, Virginia